CLINICAL TRIAL: NCT02277379
Title: Prediction of Bleeding Outcomes / Transfusion Requirements and Assessment of Perioperative Changes in Platelet Reactivity Using Point-of-care Platelet Function Testing in Patients Undergoing Cardiac Surgery
Brief Title: Prediction of Bleeding and Transfusion Outcomes and Assessment of Perioperative Platelet Reactivity in Cardiac Surgery
Status: Completed | Type: Observational
Sponsor: University of Zagreb (Other)
Responsible Party: Principal Investigator, Petricevic Mate, M.D. , Ph.D., University of Zagreb
Other Study IDs: KBCZG8.1-14/62-2
Record Dates: First submitted 2014-10-26; First posted 2014-10-29 (Estimated); Last update posted 2015-01-09 (Estimated); Status verified 2015-01

CONDITIONS: Heart Disease
Keywords: cardiac surgery ; hemorrhage ; transfusion requirements
MeSH Terms: conditions — Heart Diseases; Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Excessive bleeding after cardiopulmonary bypass (CPB) operations remains to be a persistent problem. Antiplatelet therapy (APT) is an integral component of perioperative management in patients undergoing cardiac surgery. The impact of drug induced platelet inhibition on early postoperative bleeding extent and transfusion requirements remains difficult to predict.

In addition to, resistance to antiplatelet drugs as well as perioperative increase in platelet reactivity following CPB has been reported but this phenomenon has to be comprehensively investigated.

The best point-of-care platelet function test to predict bleeding complications/transfusion requirements remains unclear. In addition to, the best test platelet function test to monitor resistance to antiplatelet therapy and its impact on clinical outcomes remains elusive.

The aim of this study is:

1. to compare two point-of-care platelet function analyzers (Multiplate and ROTEM Platelet) in regard to prediction of bleeding complications/trasfusion requirements.
2. to compare two point-of-care platelet function analyzers (Multiplate and ROTEM Platelet) in regard to detection of high "on-treatment" platelet reactivity both pre- and postoperatively.

DETAILED DESCRIPTION:
Excessive bleeding after cardiopulmonary bypass (CPB) operations remains to be a persistent problem. Antiplatelet therapy (APT) is an integral component of perioperative management in patients undergoing cardiac surgery. The impact of drug induced platelet inhibition on early postoperative bleeding extent and transfusion requirements remains difficult to predict.

In addition to, resistance to antiplatelet drugs as well as perioperative increase in platelet reactivity following CPB has been reported but this phenomenon has to be comprehensively investigated.

The best point-of-care platelet function test to predict bleeding complications/transfusion requirements remains unclear. In addition to, the best test platelet function test to monitor resistance to antiplatelet therapy and its impact on clinical outcomes remains elusive.

The aim of this study is:

1. to compare two point-of-care platelet function analyzers (Multiplate and ROTEM Platelet) in regard to prediction of bleeding complications/trasfusion requirements.

   Three different tests will be performed on each device simultaneously at three time points:

   T1) Preoperative testing will include ASPI test, ADP test and TRAP test for Multiplate device and ARATEM, ADPTEM and TRAPTEM for ROTEM Platelet device, respectively.

   T2) After declamping of the aorta: ASPI test, ADP test and TRAP test for Multiplate device and ARATEM, ADPTEM and TRAPTEM for ROTEM Platelet device will be performed.

   T3) 5-10 minutes after protamine administration: ASPI test, ADP test and TRAP test for Multiplate device and ARATEM, ADPTEM and TRAPTEM for ROTEM Platelet device will be performed.

   Results obtained with this two platelet function point-of-care devices at the first three timepoints will be tested for correlations with postoperative bleeding amount and intra/postoperative transfusion requirements. Predictibalility of bleeding complications as well as transfusion requirements will be compared between Multiplate tests and ROTEM Platelet tests.
2. to compare two point-of-care platelet function analyzers (Multiplate and ROTEM Platelet) in regard to detection of high "on-treatment" platelet reactivity both pre- and postoperatively.

To compare Multiplate and ROTEM Platelet for assessment of high on treatment platelet reactivity we will use tests being performed preoperatively (T1) and tests performed at fourth postoperative day (T4).

ASPI test (Multiplate) and ARATEM test (ROTEM Platelet) are sensitive to the platelet inhibitory effect of acetylsalicylic acid. Thus, the incidence of resistance to acetylsalicylic acid , measured by Multiplate ASPI test and ROTEM Platelet ARATEM will be compared between device measurements performed at T1 and T4, respectively. Specific subanalysis will be performed for ARATEM test with aim to make laboratory based definition of resistance to acetylsalicylic acid. Specific cut-of value for acetylsalicylic acid resistance has already been defined by our working group for Multiplate ASPI test.

ADP test (Multiplate) and ADPTEM test (ROTEM Platelet) are sensitive to the effect of thienopyridines. For patients being preoperatively exposed to thienopyridines, measurements of Multiplate ADP test and ROTEM Platelet ADPTEM test will be performed at T1 with aim to compare the incidence of high on-treatment platelet reactivity.

Preoperative (T1) and postoperative (T4) measurements obtained with Multiplate and ROTEM Platelet will be compared. Perioperative increase in platelet reactivity will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. > 18 years old
2. Elective cardiac surgery patients
3. Coronary artery disease
4. Aortic valve disease
5. Mitral valve disease
6. Ascendent aorta aneurysm
7. Combine coronary and valve disease
8. Cardiac surgery procedures using cardiopulmonary bypass

Exclusion Criteria:

1. Missing consent
2. Patients with emergent cardiac surgical procedures
3. Patients on antiplatelet therapy other than aspirin , clopidogrel and prasugrel
4. Patients with inaccurate antiplatelet therapy administration documentation
5. Missing data
6. Off-pump procedures
7. Patients younger than 18 years old
8. Patients with severe mental disorders
9. Intrinsic coagulopathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients undergoing elective cardiac surgery procedures will be consecutively enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 113 (Actual)
Dates: Start 2014-09; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
postoperative chest tube output | the first 24 postoperative hours
  Chest tube output (CTO) was determined as study's primary outcome. To estimate blood loss, we will meticulously document CTO, in first 24 postoperative hours and divide it by patient's weight. Drainage loss will be assessed after completion of a 30-minute stabilization period. Blood loss during the stabilization period will not be included in the definition of postoperative hemorrhage. Such loss may be caused by postural changes when transferring the patient from the operating room table to the bed or because of fluid in the pleural or mediastinal cavity, which may have arisen from the rinsing with water as an attempt to achieve surgical hemostasis.

SECONDARY OUTCOMES:
Transfusion requirements | 5 days
  Intraoperative and postoperative transfusion requirements (packed red blood cells in mL, fresh frozen plasma in mL, fibrinogen concentrate in grams and platelet concentrates in units) will be determined as study's secondary outcome.
reexploration for bleeding | 3 days
  Surgical reexploration of the mediastinum for excessive bleeding will be noted, along with any surgical explanation for the bleeding.

OTHER OUTCOMES:
30 day mortality | 30 day
  Patient follow up will be performed regularly as a part of a clinical routine protocol. The occurence of mortality within 30 day will be noted

CONTACTS AND LOCATIONS:
Overall Officials: Mate Petricevic, M.D., Ph.D., Principal Investigator — Clinical Hospital Centre Zagreb
Locations (1):
- UHC Zagreb, Zagreb, Croatia